CLINICAL TRIAL: NCT06260878
Title: Short-term Intravenous Fluids for Prevention of Post-ERCP Pancreatitis
Acronym: STRIPE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REB23-0625
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-02

CONDITIONS: Post-ERCP Acute Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Ringer's lactate 2500 cc IV (Experimental)
  Interventions: Other: Intravenous Ringer's lactate
- Ringer's lactate 2000 cc IV (Experimental)
  Interventions: Other: Intravenous Ringer's lactate
- Ringer's lactate 1500 cc IV (Experimental)
  Interventions: Other: Intravenous Ringer's lactate
- Ringer's lactate 1000 cc IV (Experimental)
  Interventions: Other: Intravenous Ringer's lactate
- Ringer's lactate 500 cc IV (Active Comparator)
  Interventions: Other: Intravenous Ringer's lactate

INTERVENTIONS:
Other: Intravenous Ringer's lactate — Intravenous Ringer's lactate

SUMMARY:
This study will explore the efficacies of several practical short-term (peri-procedural) intravenous fluid regimens in the prevention of post- endoscopic retrograde cholangiopancreatography (ERCP) pancreatitis (PEP). PEP is the most common serious ERCP-related adverse event (AE), occurring in 5-15% of patients, and associated with significant morbidity, mortality, and healthcare utilization. Given the current lack of data on effectiveness of short-term fluid regimens in PEP prevention to inform practice, the results of the proposed study have the strong potential to impact ERCP practices worldwide, whether positive or negative.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years (due to higher likelihood of undiagnosed cardiac disease or renal insufficiency in patients >75 years of age)
2. ability to give informed consent
3. native major papillary anatomy
4. ability and willingness to obtain bloodwork the day after ERCP

Exclusion Criteria:

1. prior ERCP with sphincterotomy and/or sphincteroplasty
2. confirmed or suspected cholangitis or sepsis
3. confirmed pancreatitis, hyperlipasemia, or hyperamylasemia within the preceding 7 days
4. NYHA Class II or greater heart failure
5. active pulmonary edema
6. myocardial infarction or ischemia within the preceding 3 months
7. renal insufficiency with CrCl < 40 mL/minute
8. CPT Class B or C cirrhosis and/or end-stage liver disease
9. room air oxygen saturation <90% or requirement of home O2
10. hypernatremia with Na+ ≥ 150 mEq/L or Na+ <130 mEq/L
11. uncontrolled hypertension or hypotension
12. pregnant status

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 505 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Serum amylase | 24 hours

SECONDARY OUTCOMES:
Pancreatitis | 7 days
  Abdominal pain characteristic of pancreatitis occurring after ERCP resulting in admission of (or prolongation of admission by) at least 2 nights, with one or more of: (1) amylase and/or lipase > 3 times the upper limit of normal when measured at least the day after ERCP and/or (2) imaging findings characteristic of pancreatitis.
Bleeding | 30 days
  Hematemesis, melena, or hematochezia (other than blood on toilet paper) resulting in one or more of the following: (1) hemoglobin drop > 2g and/or a need for transfusion, (2) a procedure performed for evaluation of suspected bleeding, and/or (3) emergency department visit and/or admission to hospital and/or prolongation of existing admission by at least one night.
Cholangitis | 14 days
  Presentation that includes all of the following: (1) temperature < 36.0°C or > 38.0°C or white blood cell count < 4,000/L or > 10,000/L and (2) increase in bilirubin, alkaline phosphatase, or transaminases compared to pre-procedure, or, if previously normal, a rise in any parameter to > 1.5 times the upper limit of normal, and (3) emergency department visit and/or admission to hospital and/or prolongation of existing admission by at least one night.
Cardiorespiratory adverse event | 7 days
  Cardiorespiratory signs and/or symptoms related to a non-gastrointestinal organ system, or sedation- or drug-related reaction occurring during or after ERCP. The event must (1) result in an unplanned emergency department visit, hospital admission, or prolongation of existing admission by at least one night and/or (2) prevent completion of the planned procedure and/or (3) result in death.
Serum lipase | 24 hours
Electrolytes | 24 hours
Creatinine | 24 hours
Brain natriuretic peptide | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Peter Lougheed Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided